CLINICAL TRIAL: NCT05327400
Title: Expression and Clinical Significance of IGHD in Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Other Study IDs: NTlyh76
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-03

CONDITIONS: Gene Expression
Keywords: Pancreatic Cancer; Clinical Significance; expression; prognosis; IGHD
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Peripheral blood from pancreatic cancer patients and healthy cancer-free patients
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pancreatic cancer patients: pathologically confirmed pancreatic cancer patients
  Interventions: Other: Pathological
- healthy people: people without no neoplastic lesions and other organic diseases

INTERVENTIONS:
Other: Pathological — The pancreatic cancer cohort and the healthy cancer-free patient cohort were divided according to pathology reports
  Groups: pancreatic cancer patients

SUMMARY:
Background ： Pancreatic cancer is the most malignant tumor in the digestive system, with low level of early diagnosis and poor prognosis. There is a lack of high sensitive and specific molecular markers in the diagnosis, treatment and prognosis of pancreatic cancer.

Objective： To explore the expression of IGHD in pancreatic cancer and its correlation with clinical parameters, and to explore its prognostic value in patients with pancreatic cancer.

Methods： In this study, qRT-PCR was used to detect IGHD expression in peripheral blood. The expression of IGHD in pancreatic cancer and healthy individuals was compared. The PCR results were combined with clinical data of patients. To compare the expression of IGHD in different pancreatic cancer stages and evaluate whether IGHD expression in peripheral blood can be a potential biomarker for the diagnosis of pancreatic cancer, chi-square test was used to analyze the factors influencing the expression level of IGHD. Kaplan-Meier was used to analyze patient prognosis, and further Cox regression analysis was used to analyze the factors influencing patient prognosis and independent risk factors.

DETAILED DESCRIPTION:
Methods：The expressions of IGHD in peripheral blood of about 30 patients with pancreatic cancer and more than 30 healthy controls were detected by qRT-PCR, and the differences of IGHD were analyzed.The expression of IGHD in pancreatic cancer and healthy individuals was compared. The PCR results were combined with clinical data of patients. To compare the expression of IGHD in different pancreatic cancer stages and evaluate whether IGHD expression in peripheral blood can be a potential biomarker for the diagnosis of pancreatic cancer, chi-square test was used to analyze the factors influencing the expression level of IGHD. Kaplan-Meier was used to analyze patient prognosis, and further Cox regression analysis was used to analyze the factors influencing patient prognosis and independent risk factors.

Pancreatic cancer is a disease of digestive system with a high degree of malignancy. The level of early diagnosis and therapeutic effect are limited by the research status of pancreatic adenocarcinoma. Conventional CT, MRI and other methods have a limited level of early diagnosis of pancreatic cancer, and EUS and endoscope-guided needle biopsy are in the stage of clinical trials. Studies on novel markers involve protein, miRNA, exosome, methylation, protein and genomics, but there is no mature and practical diagnostic method. Based on the current diagnosis, treatment and prognosis level of pancreatic cancer, I made a bold attempt to study the expression of IGHD in pancreatic cancer and their relationship with clinical parameters and prognosis level, so as to screen molecular markers conducive to diagnosis, treatment and prognosis of pancreatic cancer and provide data support for improving the diagnosis and treatment level of pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed pancreatic cancer

Exclusion Criteria:

* noperable patients
* other malignant tumors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with operable pancreatic cancer without other malignancies
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
High expression of IGHD is independent risk factors for poor prognosis in patients with pancreatic cancer. | 2022.4-2023.10
  IGHD was highly expressed in pancreatic cancer patients , but low in the healthy cancer-free patients.
  Patients with high expression of IGHD had lower prognosis. High expression of IGHD, T stage (T3T4), lymphatic metastasis and distant metastasis are independent risk factors for poor prognosis in patients with pancreatic cancer.
  Expression level of IGHD in peripheral blood cells is a potential biomarker for the diagnosis of pancreatic cancer

CONTACTS AND LOCATIONS:
Overall Officials: Lu Y Yuhua, phd, Study Director — The Affiliated Hospital of Nantong University; Chen Q Qiyang, master, Principal Investigator — Nantong University
Locations (1):
- The Affiliated Hospital of Nantong University, Nantong, Jiangsu, China